CLINICAL TRIAL: NCT03143478
Title: Mechanical Muscle Activity With Real-time Kinematics (M-MARK): A Novel Combination of Existing Technologies to Improve Arm Recovery Following Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southampton (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Imperial College London (Other); Maddison Ltd (Other); Tactiq Ltd (Unknown); University of Maryland (Other); North Bristol NHS Trust (Other); Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 01
Record Dates: First submitted 2017-04-25; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- M-MARK (Experimental): Participants self administer rehabilitation exercises using the M-MARK device for 20 days.
  Interventions: Device: M-MARK

INTERVENTIONS:
Device: M-MARK — M-MARK will be used by therapists for assessment of the upper limb, and stroke participants will be asked to use M-MARK whilst performing individually tailored and prescribed exercises for a minimum of 5 days/week.
  A set of tailored arm exercises using M-MARK (including targets for repetitive and functional activities) will be prescribed which the participant will be asked to practice independently at home for four weeks.
  During the four weeks, the patient (with support from their carer as required) will be encouraged to don the M-Mark garment and log-on to the M-Mark computer tablet each day to carry out their programme of exercises. They will be asked to use M-Mark to repeat as many exercise sessions per day as prescribed to them by their research therapist.

SUMMARY:
About 150,000 people in the UK suffer a stroke each year and ~60% with moderate to severe stroke fail to recover arm or hand use. Stroke rehabilitation is increasingly home-based following early supported discharge (ESD) from hospital to facilitate self-management and avoid problems associated with prolonged hospital stays. There is strong evidence that intensive practice and re-education of normal movement is essential for functional motor recovery, hence the NHS guideline of 45 minutes therapy 5 days per week, but NHS Trusts have difficulty meeting this target due to cost and access to specialist therapists.

An M-MARK Mk1 device that combines an Inertial Measurement Unit (IMU) with an Mechanomyography (MMG) sensor has been designed and laboratory tested. Novel signal processing techniques have been demonstrated that reduce problems of vibration artifacts and generate information on mechanical muscle activity and movement. The aim of the overall M-MARK project is to develop a low-cost wearable wireless device (Mk2) that patients can use independently at home while practicing standardised everyday activities to regain upper limb function. Mk2 M-MARK has now been developed in collaboration with therapists, patients and their carers. The system incorporates feedback, presented on a computer/tablet, as motivating visualisations of movement showing them if they have moved in the correct way. A separate interface has been developed for therapists, which offers a simple system to diagnose specific movement problems to inform clinical decision-making, monitor progress and thus increase efficiency of therapy.

In phase 1 of this study, user requirements were assessed to inform the development of the Mk2 M-MARK for clinical use. Ten patients and carers were interviewed and 20 health professionals took part in two focus groups, from Portsmouth Hospitals NHS trust and North Bristol NHS Trust. The Mk2 system has now been developed, reliability demonstrated and iterative testing with stroke patients has ensured usability of the system.

This phase of research will examine the clinical feasibility of using Mk2 M-MARK with stroke patients who are undergoing early supported discharge. All feasibility aspects of the wearable system will be assessed including usability and safety. Preliminary data on efficacy will be collected and a health economics analysis will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or older.
* Between 1 and 20 weeks post clinical diagnosis of stroke with residual upper limb movement deficits.
* Currently undergoing upper limb rehabilitation post-stroke within early supported discharge.
* Be able to lift hemiparetic arm from lap onto a table.
* Physically and cognitively able to comply with study protocol (Score 19 or higher on the Montreal cognitive assessment [9] (scores between 19-25 corresponds to mild cognitive impairment, and 25-30 represent normal cognition). For aphasic patients, the Oxford cognitive screen (OCS) will be used to determine cognitive status.
* Able to walk to or transfer to a chair and bring it up to a table nearby, independently or have assistance of a carer as required.
* Able to effectively don and doff the garment independently or have a carer who is able and willing to assist them.
* Be medically stable enough to undergo arm rehabilitation, as determined by the ESD team.

Exclusion Criteria:

* Unable to understand the purpose of the study, follow simple instructions and give informed consent
* Unable to provide useful feedback (either patient or carer) due to communication difficulties post stroke.
* A maximum level of arm function - full movement of the elbow, shoulder and hand with the only unresolved impairment being fine dexterity.
* Requirement of an interpreter.
* A skin disease or allergy to garment material including: Nylon, Polypropylene or Polyester.
* Severe pain of the hemiparetic arm, shoulder or hand, either at rest or during movement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
Movement and muscle activity parameters measured by the M-MARK system | Baseline - 4 weeks
  Kinematic and Muscle activity data recorded within the system

SECONDARY OUTCOMES:
Streamlined Wolf Motor Function Test | Baseline - 4 weeks
  Valid and reliable upper limb functional assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jane Burridge, Principal Investigator — University of Southampton

IPD SHARING:
Plan to Share IPD: No